CLINICAL TRIAL: NCT03190694
Title: A Study to Assess the Renoprotective Effects of the SGLT2 Inhibitor Dapagliflozin in Non-Diabetic Patients With Proteinuria: a Randomized Double Blind 6-Weeks Cross-Over Trial
Brief Title: Effects of Dapagliflozin in Non-diabetic Patients With Proteinuria
Acronym: DIAMOND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hiddo Lambers Heerspink (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Hiddo Lambers Heerspink, Clinical Pharmacologist, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2017003001; 2017-001090-16 (EudraCT Number)
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Diseases; Proteinuria
Keywords: chronic kidney disease; non diabetic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: A Randomized Double Blind 6-Weeks Cross-over
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 10mg Tablet, then Placebo (Experimental): Participants first received Dapagliflozin 10mg tablet for 6 weeks. After a washout period of 6 weeks, they then received Placebo tablet for 6 weeks (matching Dapagliflozin 10mg).
  Dapagliflozin 10 mg: Green, plain, diamond shaped, film coated tablet (orally) Placebo: Green, plain, diamond shaped, film coated tablet. Does not contain active ingredient
  Interventions: Drug: Dapagliflozin 10mg
- Placebo, then Dapagliflozin (Placebo Comparator): Participants first received Placebo tablet for 6 weeks. After a washout period of 6 weeks, they then received Dapagliflozin 10mg tablet for 6 weeks (matching Dapagliflozin 10mg).
  Placebo: Green, plain, diamond shaped, film coated tablet. Does not contain active ingrediënt Dapagliflozin 10 mg: Green, plain, diamond shaped, film coated tablet (orally)
  Interventions: Drug: Dapagliflozin 10mg

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Tablet
  Other Names: Placebo Matching Dapagliflozin 10mg

SUMMARY:
This study tests the hypothesis that dapagliflozin lowers proteinuria in patients with non-diabetic chronic kidney disease.

DETAILED DESCRIPTION:
Despite optimal treatment with renin-angiotensin-aldosterone-system (RAAS) inhibitors, many patients with non-diabetic kidney disease show progressive kidney function loss, which is associated with high residual proteinuria. Novel treatment strategies are therefore required to further decrease proteinuria and to slow kidney function decline.

Dapagliflozin is a sodium-glucose transport (SGLT2) inhibitor and inhibits the reabsorption of glucose and sodium in the proximal tubule. The increased natriuresis following dapagliflozin administration normalizes tubuloglomerular feedback resulting in a reduction in intra-glomerular hypertension, which is in turn manifested by acute reversible reductions in glomerular filtration rate and albuminuria. Since many etiologies of non-diabetic nephropathy are characterized by intraglomerular hypertension, we hypothesize that dapagliflozin acutely decreases GFR and proteinuria in patients without diabetes at risk of progressive kidney function loss via a glucose independent hemodynamic mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years
* Urinary protein excretion > 500 mg/g and ≤ 3500 mg/g in a 24-hr urine collection eGFR ≥ 25 mL/min/1.73m2
* On a stable dose of an ACEi or ARB for at least 4 weeks prior to randomization
* Willing to sign informed consent
* Women of Child-Bearing Potential (WOCBP):
* WOCBP must be using an acceptable method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the last dose of study drug in such a manner that the risk of pregnancy is minimized.
* WOCBP must have a negative serum or urine pregnancy test result (minimum sensitivity 25 IU/L or equivalent units of HCG) within 0 to 72 hours before the first dose of study drug.
* Women must not be breast-feeding.

WOCBP comprises women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who are not post-menopausal.

Exclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes mellitus
* Urinary protein excretion > 3500 mg/day
* Peripheral Vascular Disease
* Autosomal dominant polycystic kidney disease or autosomal recessive polycystic kidney disease, lupus nephritis, or ANCA-associated vasculitis
* Indication for immunosuppressants as per the treating physician's judgment.
* Receiving cytotoxic therapy, immunosuppressive therapy, or other immunotherapy for primary or secondary renal disease within 6 months prior to enrolment.
* Active malignancy aside from treated squamous cell or basal cell carcinoma of the skin.
* Use of co-interventional treatments (outlined in section 4.2 of the protocol) within 6 weeks of screening will not be allowed.
* Any medication, surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of medications including, but not limited to any of the following:

  * History of active inflammatory bowel disease within the last six months;
  * Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  * Gastro-intestinal ulcers and/or gastrointestinal or rectal bleeding within last six months;
  * Pancreatic injury or pancreatitis within the last six months;
  * Evidence of hepatic disease as determined by any one of the following: ALT or AST values exceeding 3x ULN at the screening visit, a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt;
  * Evidence of urinary obstruction of difficulty in voiding at screening
* History of severe hypersensitivity or contraindications to dapagliflozin
* Subject who, in the assessment of the investigator, may be at risk for dehydration or volume depletion that may affect the interpretation of efficacy or safety data
* Participation in any clinical investigation within 3 months prior to initial dosing.
* Donation or loss of 400 ml or more of blood within 8 weeks prior to initial dosing.
* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* Pregnancy or breastfeeding
* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and up to 4 weeks after the last dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-11-12 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (2):
  - Nephrology Dept., Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - Division of Nephrology University Health Network, University of Toronto, Toronto, Ontario
- Malaysia (2):
  - Nephrology Unit, University Kebangsaan Malaysia, Kuala Lumpur
  - University Malaya Medical Centre, Ward 8TE, Kuala Lumpur
- Netherlands (3):
  - Dept Internal Medicine, division of Nephrology Hospital Group Twente, Almelo
  - Dept.of Nephrology, VU University Medical Center, Amsterdam
  - Dept. Nephrology, University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Aart-van der Beek AB, Koomen JV, Dekkers CCJ, Barbour SJ, Boulton DW, Gansevoort RT, Greasley PJ, Abdul Gafor AH, Laverman GD, Li Q, Lim SK, Stevens J, Vervloet MG, Singh S, Cattran DC, Reich HN, Cherney DZI, Heerspink HJL. Evaluation of the Pharmacokinetics and Exposure-Response Relationship of Dapagliflozin in Patients without Diabetes and with Chronic Kidney Disease. Clin Pharmacokinet. 2021 Apr;60(4):517-525. doi: 10.1007/s40262-020-00956-1. Epub 2021 Feb 15. PMID 33587286
- [Derived] Cherney DZI, Dekkers CCJ, Barbour SJ, Cattran D, Abdul Gafor AH, Greasley PJ, Laverman GD, Lim SK, Di Tanna GL, Reich HN, Vervloet MG, Wong MG, Gansevoort RT, Heerspink HJL; DIAMOND investigators. Effects of the SGLT2 inhibitor dapagliflozin on proteinuria in non-diabetic patients with chronic kidney disease (DIAMOND): a randomised, double-blind, crossover trial. Lancet Diabetes Endocrinol. 2020 Jul;8(7):582-593. doi: 10.1016/S2213-8587(20)30162-5. PMID 32559474

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then Dapagliflozin: Participants first received Placebo tablet for 6 weeks. After a washout period of 6 weeks, they then received Dapagliflozin 10mg tablet for 6 weeks.
  Placebo: Green, plain, diamond shaped, film coated tablet. Does not contain active ingredient
  Dapagliflozin 10mg: Green, plain, diamond shaped, film coated tablet (orally)
Period: Period 1
Arm/Group | Dapagliflozin 10mg Tablet, Then Placebo | Placebo, Then Dapagliflozin
Started | 27 | 26
Completed | 26 | 26
Not Completed | 1 | 0
Period: Period 2 (After 6 Weeks Wash-out)
Arm/Group | Dapagliflozin 10mg Tablet, Then Placebo | Placebo, Then Dapagliflozin
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0
Period: Wash-out and Follow-up
Arm/Group | Dapagliflozin 10mg Tablet, Then Placebo | Placebo, Then Dapagliflozin
Started | 26 | 26
Completed | 24 | 26
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dapagliflozin 10mg Tablet: 10 mg Green, plain, diamond shaped, film coated tablet (orally)
  Dapagliflozin 10mg: Tablet
- Placebo Matching Dapagliflozin Tablet: Green, plain, diamond shaped, film coated tablet. Does not contain active ingredient
  Dapagliflozin 10mg: Tablet
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10mg Tablet | Placebo Matching Dapagliflozin Tablet | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (10) | 51 (16) | 51 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 18 | 18 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asia | 11 | 6 | 17
  Hispanic | 2 | 0 | 2
  Caucasian | 12 | 17 | 29
  Other | 2 | 3 | 5
Proteinuria [Median (Inter-Quartile Range); unit: mg/24h] | 1170 [730 to 1690] | 1105 [720 to 1530] | 1110 [730 to 1560]
mGFR [Mean (Standard Deviation); unit: ml/min/1.73m2] | 58.9 (20.7) | 57.8 (25.5) | 58.3 (23.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in 24-hr Proteinuria With Dapagliflozin for Six Weeks Relative to Placebo in Patients With Non-diabetic Kidney Disease and Proteinuria 500 mg/Day on Stable Angiotensin-converting Enzyme Inhibitor or Angiotensin II Receptor Blocker Treatment.
Description: bioequivalence
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: % change from baseline
Arm/Group | Dapagliflozin 10mg Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 53 | 52
% change from baseline | -15.04 [-25.70 to -2.76] | -15.80 [-26.43 to -3.54]

2. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on Glomerular Filtration Rate (GFR) Using Iohexol Clearance
Description: bioequivalence
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: mL/min per 1.73m2
Groups:
- Dapagliflozin 10mg: Tablet: 10 mg Green, plain, diamond shaped, film coated tablet (orally)
Arm/Group | Dapagliflozin 10mg: Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 53 | 52
mL/min per 1.73m2 | -6.3 [-8.0 to -4.6] | 0.3 [-1.4 to 2.0]

3. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on Systolic/Diastolic Blood Pressure
Description: bioequivalence
Time Frame: week 0, 3, 6, 12, 15, 18, 24
Population: Due to several missed visits the no. of analyzed participants is not the same for all visits.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Dapagliflozin for 1st 6 Weeks and Matching Placebo for 6 Weeks After 6 Week Washout.: Participants first received Dapagliflozin 10mg tablet for 6 weeks. After a washout period of 6 weeks, they then received Placebo tablet for 6 weeks (matching Dapagliflozin 10mg)
- Placebo for the 1st 6 Weeks and Dapagliflozin for 6 Weeks After 6 Week Washout.: Participants first received Placebo tablet for 6 weeks. After a washout period of 6 weeks, they then received Dapagliflozin 10mg tablet for 6 weeks (matching Dapagliflozin 10mg).
Arm/Group | Dapagliflozin for 1st 6 Weeks and Matching Placebo for 6 Weeks After 6 Week Washout. | Placebo for the 1st 6 Weeks and Dapagliflozin for 6 Weeks After 6 Week Washout.
Number analyzed (Participants) | 27 | 26
mm Hg
  week 0 SBP | 127.4 (16.44) | 124.6 (13.1)
  week 3 SBP: number analyzed (Participants) | 26 | 24
  week 3 SBP | 124.3 (13.93) | 121.8 (9.9)
  week 6 SBP: number analyzed (Participants) | 26 | 26
  week 6 SBP | 120.4 (13.87) | 123.2 (12.27)
  week 12 SBP: number analyzed (Participants) | 26 | 26
  week 12 SBP | 125.6 (15.86) | 125.2 (14.02)
  week 15 SBP: number analyzed (Participants) | 25 | 24
  week 15 SBP | 125.0 (15.05) | 122.8 (13.20)
  week 18 SBP: number analyzed (Participants) | 25 | 26
  week 18 SBP | 123.5 (10.94) | 120.9 (16.48)
  week 24 SBP: number analyzed (Participants) | 24 | 26
  week 24 SBP | 123.6 (14.90) | 123.9 (14.67)
  Week 0 DBP | 77.2 (8.68) | 75.2 (7.77)
  Week 3 DBP: number analyzed (Participants) | 26 | 24
  Week 3 DBP | 78.0 (6.81) | 74.5 (6.82)
  Week 6 DBP: number analyzed (Participants) | 26 | 26
  Week 6 DBP | 74.5 (6.8) | 74.4 (7.84)
  Week 12 DBP: number analyzed (Participants) | 26 | 26
  Week 12 DBP | 77.6 (7.83) | 74.7 (9.05)
  Week 15 DBP: number analyzed (Participants) | 25 | 24
  Week 15 DBP | 77.6 (7.18) | 74.3 (8.39)
  Week 18 DBP: number analyzed (Participants) | 25 | 26
  Week 18 DBP | 76.6 (7.44) | 72.7 (9.3)
  Week 24 DBP: number analyzed (Participants) | 24 | 26
  Week 24 DBP | 74.5 (6.36) | 75.1 (8.69)

4. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on Body Weight
Description: bioequivalence
Time Frame: week 0, 3, 6, 12, 15, 18, 24
Population: Several participants missed some of their visits
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Dapagliflozin for 1st 6 Weeks and Matching Placebo for 6 Weeks After: Participants first received Dapagliflozin 10mg tablet for 6 weeks. After a washout period of 6 weeks, they then received Placebo tablet for 6 weeks (matching Dapagliflozin 10mg)
Arm/Group | Placebo for the 1st 6 Weeks and Dapagliflozin for 6 Weeks After 6 Week Washout. | Dapagliflozin for 1st 6 Weeks and Matching Placebo for 6 Weeks After
Number analyzed (Participants) | 26 | 27
kg
  Week 0 | 79.646 (15.5147) | 86.196 (23.9748)
  Week 3: number analyzed (Participants) | 24 | 26
  Week 3 | 78.892 (15.8944) | 83.242 (21.8429)
  Week 6: number analyzed (Participants) | 26 | 26
  Week 6 | 80.419 (16.1250) | 85.185 (24.2097)
  Week 12: number analyzed (Participants) | 26 | 26
  Week 12 | 78.712 (15.0825) | 85.265 (24.3126)
  Week 15: number analyzed (Participants) | 24 | 25
  Week 15 | 77.046 (15.1826) | 83.048 (22.8179)
  Week 18: number analyzed (Participants) | 26 | 25
  Week 18 | 77.488 (14.9676) | 86.144 (24.4698)
  Week 24: number analyzed (Participants) | 23 | 24
  Week 24 | 77.204 (12.4649) | 84.163 (22.2775)

5. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on 6-keto-Prostaglandin F1 Alpha/Creatinine Ratio
Description: bioequivalence
Time Frame: Baseline, Week 6
Population: Difference in no. of participants at week 6 due to missed visit
Measure: Mean (Standard Deviation); unit: pg/mmol
Groups:
- Dapagliflozin 10mg: Tablet: 0 mg Green, plain, diamond shaped, film coated tablet (orally)
Arm/Group | Dapagliflozin 10mg: Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 51 | 50
pg/mmol
  Baseline | 0.1170 (0.0422) | 0.1167 (0.1079)
  Week 6: number analyzed (Participants) | 50 | 50
  Week 6 | 0.1281 (0.0450) | 0.1203 (0.0554)

6. Secondary Outcome: Safety of Dapagliflozin vs. Placebo - the Number of Participatns With Hypoglycemic Events and/or Serious Adverse Events
Description: safety
Time Frame: week 0-26
Measure: Number; unit: participants
Arm/Group | Dapagliflozin 10mg Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 53 | 52
participants
  Hypoglycemic episode | 0 | 0
  Serious adverse event | 1 | 1

7. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on Adenosine/Creatinine Ratio
Description: bioequivalence
Time Frame: Baseline, Week 6
Population: Difference in no. of participants at week 6 due to missed visit
Measure: Mean (Standard Deviation); unit: micromol/mmol
Arm/Group | Dapagliflozin 10mg: Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 51 | 50
micromol/mmol
  Baseline | 0.2020 (0.1566) | 0.1949 (0.1529)
  Week 6 | 0.2218 (0.1706) | 0.2373 (0.2529)

8. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on Prostaglandin E2/Creatinine Ratio
Description: bioequivalence
Time Frame: Baseline, Week 6
Population: Difference in no. of participants at week 6 due to missed visit
Measure: Mean (Standard Deviation); unit: pg/mmol
Arm/Group | Dapagliflozin 10mg: Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 51 | 50
pg/mmol
  Baseline | 0.1131 (0.1498) | 0.0980 (0.1034)
  Week 6 | 0.1702 (0.2656) | 0.0946 (0.1428)

9. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on Thromboxane B2/Creatinine Ratio
Description: bioequivalence
Time Frame: Baseline, Week 6
Population: Difference in no. of participants at week 6 due to missed visit
Measure: Mean (Standard Deviation); unit: pg/mmol
Arm/Group | Dapagliflozin 10mg: Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 51 | 50
pg/mmol
  Baseline | 0.0921 (0.0569) | 0.0963 (0.0470)
  Week 6 | 0.1058 (0.1005) | 0.0930 (0.0499)

10. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on PGEM/Creatinine Ratio
Description: bioequivalence
Time Frame: Baseline, Week 6
Population: Difference in no. of participants at week 6 due to missed visit
Measure: Mean (Standard Deviation); unit: pg/mmol
Arm/Group | Dapagliflozin 10mg: Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 51 | 50
pg/mmol
  Baseline | 0.0989 (0.0559) | 0.0948 (0.0552)
  Week 6: number analyzed (Participants) | 50 | 50
  Week 6 | 0.0965 (0.0538) | 0.0963 (0.0565)

11. Secondary Outcome: Effect of Dapagliflozin 10 mg/d Compared to Placebo on NTproBNP
Description: bioequivalence
Time Frame: Baseline (week 0, week 12), Week 6 + 18 (pooled)
Population: Difference in no. of participants at week 6 due to missed visit
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Dapagliflozin 10mg: Tablet | Placebo Matching Dapagliflozin Tablet
Number analyzed (Participants) | 52 | 50
ng/L
  Baseline (week 0 + 12) | 118.8 (151.18) | 125.0 (161.10)
  Week 6 + 18: number analyzed (Participants) | 51 | 50
  Week 6 + 18 | 108.7 (148.74) | 152.6 (277.74)

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent and throughout the study, including the run-in and wash-out periods, until the follow-up visit 6 weeks after the last treatment period.
Arm/Group | Dapagliflozin 10mg Tablet | Placebo Matching Dapagliflozin Tablet
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/52
Other Adverse Events (participants affected / at risk) | 17/53 | 13/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg Tablet (N=53) | Placebo Matching Dapagliflozin Tablet (N=52)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Colon Cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg Tablet (N=53) | Placebo Matching Dapagliflozin Tablet (N=52)
Any adverse event (General disorders) | 17 (17) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT03190694/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03190694/SAP_001.pdf